CLINICAL TRIAL: NCT07069010
Title: Evaluation of Burnout Syndrome Among Healthcare Professionals in Intensive Care Units Within the EPIC (Enhancing Palliative Care in ICU) Research
Brief Title: Burnout Syndrome in the Intensive Care Unit Before and During a Palliative Care Trial
Acronym: BURNOUT-EPIC
Status: Recruiting | Type: Observational
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Spyros D. Mentzelopoulos, Professor in Intensive Care Medicine, National and Kapodistrian University of Athens Medical School, University of Athens
Other Study IDs: 247-24/4/2024
Record Dates: First submitted 2025-07-07; First posted 2025-07-16 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Burnout Syndrome
Keywords: ICU burnout; Moral distress; self compassion; Tele-palliative care; repeated measures survey
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ICU healthcare professionals

SUMMARY:
One hundred ICU doctors, nurses and psychologists from the 28 units participating in the EPIC stepped-wedge trial (ClinicalTrials.gov NCT06605079) will each complete the same four-part survey twice-once during their unit's usual-care phase and again during the EPIC tele-palliative-care intervention. The questionnaire begins with Part A, gathering demographic and professional details such as age, gender, family status, education, role, years of ICU service, shift patterns, leave days and any prior palliative-care or ethics training. Part B then probes 22 workplace stressors and ethical dilemmas-resource constraints, family pressures, moral conflicts, emotional distancing from colleagues, perceived control over decisions and work-life balance-using a five-point frequency scale. Part C merges a 19-item Maslach Burnout Inventory subset (emotional exhaustion, depersonalization, personal accomplishment) on a seven-point frequency scale with a 16-item Oldenburg Burnout Inventory subset (exhaustion, disengagement) on a four-point agreement scale. Finally, Part D employs Neff's 16-item Self-Compassion Scale-rated from almost never to almost always-to assess self-kindness, common humanity, mindfulness, self-judgment, isolation and over-identification. Within-subject, repeated-measures analyses of total and subscale scores will quantify how EPIC's blended-learning curriculum and standardized teleconsultations shift clinician burnout profiles and self-compassion over time.

DETAILED DESCRIPTION:
One hundred ICU physicians, nurses and clinical psychologists drawn from the twenty-eight adult units enrolled in the EPIC stepped-wedge trial (ClinicalTrials.gov NCT06605079) will each complete an identical four-part survey twice-once during their unit's usual-care phase and again after crossover into the EPIC tele-palliative-care intervention. Administered in two stages (Parts A and B via secure email link; Parts C and D during a facilitated online session), the entire battery requires about forty minutes per administration and produces detailed profiles of clinician demographics, workplace stressors, core burnout dimensions and self-compassion. Within-subject repeated-measures analyses will then quantify how the combination of blended-learning palliative-care modules and standardized teleconsultations influences individual well-being over time.

Part A consists of fifteen fixed-response items capturing demographic and professional background. Respondents select from categorical options for gender (male/female), age bracket, family status and number of children, as well as highest educational attainment (secondary, vocational, undergraduate, postgraduate, PhD) and whether they have previously received palliative-care or ethics training (yes/no). Work-related variables include role (doctor, nurse, psychologist), years of ICU experience (0-10, 10-20, 20-30, >30), average evening hours per month (<3, 3-5, >5), typical nightly sleep duration (<5 hours, 5-7 hours, >7 hours) and annual leave days (<15, 15-30, >30). Participants also indicate the type of unit in which they work (mixed/multi-purpose, surgical, cardiology or other). These objective data provide essential covariates for exploring whether baseline characteristics moderate the EPIC intervention's effects on burnout and self-compassion trajectories.

Part B probes the frequency of twenty-two common ICU stressors and ethical dilemmas using a five-point Likert frequency scale (1 = Never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Always). Questions address emotional distance from colleagues, resource constraints that force care adjustments, pressure from patient families, internal moral conflict between life-support and quality-of-life decisions, perceived control over treatment choices, work-life balance and opportunities for professional development. For example, clinicians rate how often they must limit treatments due to limited resources, experience doubts about ethical issues in prognostic decision-making or feel that their performance does not reflect their skills. By capturing both external pressures and internal moral distress, Part B establishes a baseline against which EPIC's specialist palliative consultations can be assessed for stress-reduction efficacy.

Part C combines two respected burnout instruments. The first is a nineteen-item subset of the Maslach Burnout Inventory (MBI), administered on a seven-point frequency scale (1 = Never, 2 = A few times a year, 3 = Once a month, 4 = A few times a month, 5 = Once a week, 6 = A few times a week, 7 = Every day). Items form three subscales-emotional exhaustion (for instance, "I feel emotionally drained by my work"), depersonalization ("I treat some patients as if they were objects") and personal accomplishment ("I feel I have achieved many worthwhile things in this job"). Previous ICU studies consistently report Cronbach's alpha of approximately 0.90 for the MBI total and its subscales, indicating excellent internal consistency. The second is a sixteen-item subset of the Oldenburg Burnout Inventory (OLBI), using a four-point agreement scale (1 = Strongly agree, 2 = Probably agree, 3 = Probably disagree, 4 = Strongly disagree). The OLBI yields two subscales-exhaustion ("After work I often feel worn out") and disengagement ("I feel indifferent toward my work"). Cronbach's alpha for the combined OLBI scale typically exceeds 0.80, with subscale values around 0.87 for exhaustion and 0.81 for disengagement. By utilizing both instruments, Part C captures affective depletion and cognitive withdrawal components of burnout, providing a comprehensive measurement of clinicians' occupational distress.

Part D employs the full sixteen-item Self-Compassion Scale developed by Neff, rated on a five-point frequency scale (1 = Almost never, 2 = Rarely, 3 = Sometimes, 4 = Often, 5 = Almost always). Items evaluate three positive dimensions-self-kindness, common humanity and mindfulness-and their negative counterparts-self-judgment, isolation and over-identification. Sample statements include "I try to be understanding toward those aspects of my personality I don't like" and "When I'm feeling down I tend to obsess on everything that's wrong." In Greek ICU populations, both the positive and negative subscales consistently achieve Cronbach's alpha near 0.86, confirming reliable assessment of clinicians' self-compassion levels. Because higher self-compassion has been shown to buffer against burnout, Part D provides critical insight into personal resilience factors that EPIC may enhance.

To maximize data integrity, Parts A and B are distributed seven days before the scheduled online session via encrypted email links, allowing clinicians to complete demographic and stressor items thoughtfully at their convenience. During a facilitator-led videoconference, respondents then complete Parts C and D in real time, with on-screen guidance to clarify any item interpretations. Electronic responses are pseudonymized and stored in a secure database meeting GDPR requirements. Ethical approval covers both survey administrations, and informed consent materials emphasize voluntary participation, the right to withdraw at any point and assurances that individual responses will remain confidential and not influence professional evaluations.

The primary analytical objective is to test within-subject changes in total and subscale scores for Part B stressors, Part C burnout dimensions and Part D self-compassion between the control and EPIC phases. Mixed-effects models-with clinician as a random intercept and fixed effects for time period, unit and relevant Part A covariates such as years of experience or prior palliative training-will assess whether the blended-learning modules and teleconsultations yield statistically significant reductions in emotional exhaustion, depersonalization and disengagement, alongside increases in self-compassion. Secondary analyses will explore moderation by baseline characteristics, clarifying which clinician subgroups derive the greatest benefit from EPIC. Effect sizes will be interpreted against established benchmarks for within-subject interventions, with special attention to medium-sized shifts in Cronbach's alpha-validated scales.

By integrating rich background profiles, a granular inventory of ICU stressors, complementary burnout measures and a validated self-compassion assessment-all framed within a robust repeated-measures design-this extended four-part survey promises nuanced insights into how telemedicine-enabled palliative-care integration can bolster resilience, reduce moral distress and foster sustainable clinician engagement in the high-pressure ICU environment.

Sample Size Determination A priori power analysis using a one-group, two-measurement repeated-measures ANOVA (within-subjects) indicated that, to detect a medium effect size (f = 0.25) on the primary outcome (within-subject change in composite burnout score) with α = 0.01, 95% power, a correlation of 0.5 between pre- and during-intervention scores, and perfect sphericity (ε = 1), 75 clinicians are required (denominator df = 74, λ = 18.75, critical F = 6.99). To allow for up to 25% attrition and support subgroup and moderator analyses, the target enrollment is set at 100 ICU clinicians.

Multivariable mixed-effects logistic regression will test the odds of a clinically meaningful burnout change-defined by 95% minimal detectable change thresholds (≥7-point reduction on the Maslach Burnout Inventory or ≥8-point reduction on the Oldenburg Burnout Inventory). The binary responder outcome (achieved vs. not achieved) will include a random intercept for ICU site to account for clustering.

Fixed-effect predictors (up to 10) will include:

* Age (years)
* Gender
* Profession (nurse, physician, other)
* Years of ICU experience
* Unit type (medical, surgical, mixed)
* Shift pattern (day, night, mixed)
* Baseline burnout score
* Baseline self-compassion score
* Prior palliative-care training (yes/no)
* EPIC trial phase (intervention vs. control)

ELIGIBILITY:
Inclusion Criteria:

* ICU clinicians (nurses, physicians, advanced practice providers) actively caring for critically ill patients
* Employed in participating ICUs for ≥3 months prior to study start
* Willing to complete both pre- and during-intervention surveys
* Consent to participate in educational tele-palliative care trial

Exclusion Criteria:

* Locum tenens or temporary staff not continuously assigned to the unit
* Clinicians on leave (medical, parental, or extended leave) during either survey period
* Prior enrollment in similar palliative care training within past 6 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study will enroll ~100 multidisciplinary ICU clinicians-staff physicians, registered nurses and advanced practice providers-who have been continuously assigned to participating adult intensive care units for at least three months prior to study start. All participants will complete Greek-language pre- and during-intervention psychometric surveys and engage in the tele-palliative care educational intervention. Temporary or locum staff not continuously on the unit and those on leave during either survey period are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in clinician burnout by the Maslach Burnout Inventory (MBI) | 3 years
  Within-subject average percent change in clinician burnout, defined as the average of percent changes in the Emotional Exhaustion, Depersonalization and Personal Accomplishment subscores between the usual care phase and the palliative care intervention phase. Emotional Exhaustion, Depersonalization and Personal Accomplishment subscores range within 0-54, 0-30 and 0-48, respectively. Higher subscores of the first two subcomponents and lower subscore of the third subcomponent indicate worse burnout.
Change in clinician burnout by the Oldenburg Burnout Inventory (OLBI) | 3 years
  Within-subject average percent change in clinician burnout, defined as the average of percent changes in the Exhaustion and Disengagement subscores between the usual care phase and the palliative care intervention phase. Exhaustion and Disengagement subscores range within 0-32 and 0-32, respectively. Higher subscores of both subcomponents indicate worse burnout.

SECONDARY OUTCOMES:
ICU stressors and moral dilemmas frequency | 3 years
  Percent change in total frequency score and in key clusters (resource constraints, family pressures, moral conflict, emotional distancing, control, work-life balance, professional development)
Maslach Burnout Inventory subscale scores | 3 years
  Percent change in Emotional Exhaustion, Depersonalization and Personal Accomplishment subscores between the usual care phase and the palliative care intervention phase.. Emotional Exhaustion, Depersonalization and Personal Accomplishment subscores range within 0-54, 0-30 and 0-48, respectively. Higher subscores of the first two subcomponents and lower subscore of the third subcomponent indicate worse burnout.
Oldenburg Burnout Inventory subscale scores | 3 years
  Percent change in Exhaustion and Disengagement subscores between the usual care phase and the palliative care intervention phase. Exhaustion and Disengagement subscores subscores range within 0-32 and 0-32, respectively. Higher subscores of both subcomponents indicate worse burnout.
Self-Compassion Score -Short Form | 3 years
  Percent change in the short form version of Neff's self-compassion score. The self compassion score ranges within 0-5, with higher values indicating higher self compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- National and Kapodistrian University of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
Personal data protection

REFERENCES:
- [Background] White DB, Angus DC, Shields AM, Buddadhumaruk P, Pidro C, Paner C, Chaitin E, Chang CH, Pike F, Weissfeld L, Kahn JM, Darby JM, Kowinsky A, Martin S, Arnold RM; PARTNER Investigators. A Randomized Trial of a Family-Support Intervention in Intensive Care Units. N Engl J Med. 2018 Jun 21;378(25):2365-2375. doi: 10.1056/NEJMoa1802637. Epub 2018 May 23. PMID 29791247
- [Background] Weissman DE, Meier DE. Identifying patients in need of a palliative care assessment in the hospital setting: a consensus report from the Center to Advance Palliative Care. J Palliat Med. 2011 Jan;14(1):17-23. doi: 10.1089/jpm.2010.0347. Epub 2010 Dec 6. PMID 21133809
- [Background] Martin-Loeches I, De Waele JJ, Timsit JF, Bassetti M. Conventional amphotericin B must be avoided in Candida infections. Intensive Care Med. 2020 Mar;46(3):560-561. doi: 10.1007/s00134-019-05784-x. Epub 2019 Nov 29. No abstract available. PMID 31784799
- [Background] Vallbracht M, Rehwaldt S, Klupp BG, Mettenleiter TC, Fuchs W. Functional Role of N-Linked Glycosylation in Pseudorabies Virus Glycoprotein gH. J Virol. 2018 Apr 13;92(9):e00084-18. doi: 10.1128/JVI.00084-18. Print 2018 May 1. PMID 29437979
- [Background] Ubel PA, Scherr KA, Fagerlin A. Empowerment Failure: How Shortcomings in Physician Communication Unwittingly Undermine Patient Autonomy. Am J Bioeth. 2017 Nov;17(11):31-39. doi: 10.1080/15265161.2017.1378753. PMID 29111936
- [Background] Sundin EC, Horowitz MJ. Impact of Event Scale: psychometric properties. Br J Psychiatry. 2002 Mar;180:205-9. doi: 10.1192/bjp.180.3.205. PMID 11872511
- [Background] Mark NM, Rayner SG, Lee NJ, Curtis JR. Global variability in withholding and withdrawal of life-sustaining treatment in the intensive care unit: a systematic review. Intensive Care Med. 2015 Sep;41(9):1572-85. doi: 10.1007/s00134-015-3810-5. Epub 2015 Apr 23. PMID 25904183
- [Background] Barbieri JS, Frieden IJ, Nagler AR. Isotretinoin, Patient Safety, and Patient-Centered Care-Time to Reform iPLEDGE. JAMA Dermatol. 2020 Jan 1;156(1):21-22. doi: 10.1001/jamadermatol.2019.3270. No abstract available. PMID 31664426
- [Background] Song X, Liu X, Dong R, Kummer KA, Wang C. Implementation of Tele-Intensive Care Unit Services During the COVID-19 Pandemic: A Systematic Literature Review and Updated Experience from Shandong Province. Telemed J E Health. 2023 May;29(5):646-656. doi: 10.1089/tmj.2022.0302. Epub 2022 Oct 11. PMID 36251955
- [Background] From the Editor-in-Chief. Postgrad Med. 1973 Jun;53(7):25. doi: 10.1080/00325481.1973.11713476. No abstract available. PMID 27392663
- [Background] Levinson W, Kao A, Kuby A, Thisted RA. Not all patients want to participate in decision making. A national study of public preferences. J Gen Intern Med. 2005 Jun;20(6):531-5. doi: 10.1111/j.1525-1497.2005.04101.x. PMID 15987329
- [Background] Benetti F, Baldi E, Bucherelli C, Blandina P, Passani MB. Histaminergic ligands injected into the nucleus basalis magnocellularis differentially affect fear conditioning consolidation. Int J Neuropsychopharmacol. 2013 Apr;16(3):575-82. doi: 10.1017/S1461145712000181. Epub 2012 Mar 15. PMID 22418001
- [Background] Schwarzkopf D, Ruddel H, Thomas-Ruddel DO, Felfe J, Poidinger B, Matthaus-Kramer CT, Hartog CS, Bloos F. Perceived Nonbeneficial Treatment of Patients, Burnout, and Intention to Leave the Job Among ICU Nurses and Junior and Senior Physicians. Crit Care Med. 2017 Mar;45(3):e265-e273. doi: 10.1097/CCM.0000000000002081. PMID 27776092
- [Background] Schroeder DA, Stephens E, Colgan D, Hunsinger M, Rubin D, Christopher MS. A Brief Mindfulness-Based Intervention for Primary Care Physicians: A Pilot Randomized Controlled Trial. Am J Lifestyle Med. 2016 Feb 4;12(1):83-91. doi: 10.1177/1559827616629121. eCollection 2018 Jan-Feb. PMID 30202383
- [Background] Schoenherr LA, Cook A, Peck S, Humphreys J, Goto Y, Saks NT, Huddleston L, Elia G, Pantilat SZ. Proactive Identification of Palliative Care Needs Among Patients With COVID-19 in the ICU. J Pain Symptom Manage. 2020 Sep;60(3):e17-e21. doi: 10.1016/j.jpainsymman.2020.06.008. Epub 2020 Jun 14. PMID 32544647
- [Background] Scandrett KG, Reitschuler-Cross EB, Nelson L, Sanger JA, Feigon M, Boyd E, Chang CH, Paice JA, Hauser JM, Chamkin A, Balfour P, Stolbunov A, Bennett CL, Emanuel LL. Feasibility and effectiveness of the NEST13+ as a screening tool for advanced illness care needs. J Palliat Med. 2010 Feb;13(2):161-9. doi: 10.1089/jpm.2009.0170. PMID 19821699
- [Background] Aiken LH, Sloane DM, Cimiotti JP, Clarke SP, Flynn L, Seago JA, Spetz J, Smith HL. Implications of the California nurse staffing mandate for other states. Health Serv Res. 2010 Aug;45(4):904-21. doi: 10.1111/j.1475-6773.2010.01114.x. Epub 2010 Apr 9. PMID 20403061
- [Background] Raab K. Mindfulness, self-compassion, and empathy among health care professionals: a review of the literature. J Health Care Chaplain. 2014;20(3):95-108. doi: 10.1080/08854726.2014.913876. PMID 24926896
- [Background] Gomez-Veiga F, Alcaraz-Asensio A, Burgos-Revilla J, Cozar-Olmo J. Developments in urologic oncology "OncoForum": The best of 2017. Actas Urol Esp (Engl Ed). 2018 Oct;42(8):488-498. doi: 10.1016/j.acuro.2018.06.001. Epub 2018 Jun 21. English, Spanish. PMID 29935800
- [Background] Xue H, Ren C, Yang J, Sun Z, Li S, Jin Z, Shen K, Zhou W. Histogram analysis of apparent diffusion coefficient for the assessment of local aggressiveness of cervical cancer. Arch Gynecol Obstet. 2014 Aug;290(2):341-8. doi: 10.1007/s00404-014-3221-9. Epub 2014 Apr 1. PMID 24687746
- [Background] Schoener CA, Hutson HN, Peppas NA. pH-responsive hydrogels with dispersed hydrophobic nanoparticles for the oral delivery of chemotherapeutics. J Biomed Mater Res A. 2013 Aug;101(8):2229-36. doi: 10.1002/jbm.a.34532. Epub 2012 Dec 28. PMID 23281185
- [Background] Michalsen A, Neitzke G, Dutzmann J, Rogge A, Seidlein AH, Jobges S, Burchardi H, Hartog C, Nauck F, Salomon F, Duttge G, Michels G, Knochel K, Meier S, Gretenkort P, Janssens U. [Overtreatment in intensive care medicine-recognition, designation, and avoidance : Position paper of the Ethics Section of the DIVI and the Ethics section of the DGIIN]. Med Klin Intensivmed Notfmed. 2021 May;116(4):281-294. doi: 10.1007/s00063-021-00794-4. Epub 2021 Mar 1. German. PMID 33646332
- [Background] Mentzelopoulos SD, Chen S, Nates JL, Kruser JM, Hartog C, Michalsen A, Efstathiou N, Joynt GM, Lobo S, Avidan A, Sprung CL; End-of-life Practice Score Study Group. Derivation and performance of an end-of-life practice score aimed at interpreting worldwide treatment-limiting decisions in the critically ill. Crit Care. 2022 Apr 13;26(1):106. doi: 10.1186/s13054-022-03971-9. PMID 35418103
- [Background] Maslach C, Schaufeli WB, Leiter MP. Job burnout. Annu Rev Psychol. 2001;52:397-422. doi: 10.1146/annurev.psych.52.1.397. PMID 11148311
- [Background] Maslach C, Leiter MP. Understanding the burnout experience: recent research and its implications for psychiatry. World Psychiatry. 2016 Jun;15(2):103-11. doi: 10.1002/wps.20311. PMID 27265691
- [Background] Perrochon A, Kemoun G. The Walking Trail-Making Test is an early detection tool for mild cognitive impairment. Clin Interv Aging. 2014;9:111-9. doi: 10.2147/CIA.S53645. Epub 2014 Jan 7. PMID 24426778
- [Background] MacBeth A, Gumley A. Exploring compassion: a meta-analysis of the association between self-compassion and psychopathology. Clin Psychol Rev. 2012 Aug;32(6):545-52. doi: 10.1016/j.cpr.2012.06.003. Epub 2012 Jun 23. PMID 22796446
- [Background] Ma J, Chi S, Buettner B, Pollard K, Muir M, Kolekar C, Al-Hammadi N, Chen L, Kollef M, Dans M. Early Palliative Care Consultation in the Medical ICU: A Cluster Randomized Crossover Trial. Crit Care Med. 2019 Dec;47(12):1707-1715. doi: 10.1097/CCM.0000000000004016. PMID 31609772
- [Background] Oner A, Lips T, Walter U, Storch A, Ince H, Caglayan E, Yucel S, Ortak J, Schmidt C. Detection of arrhythmia using an implantable cardiac monitor following a cryptogenic stroke: a single-center observational study. Eur J Med Res. 2020 Jun 29;25(1):25. doi: 10.1186/s40001-020-00424-3. PMID 32600384
- [Background] Khandelwal N, Kross EK, Engelberg RA, Coe NB, Long AC, Curtis JR. Estimating the effect of palliative care interventions and advance care planning on ICU utilization: a systematic review. Crit Care Med. 2015 May;43(5):1102-11. doi: 10.1097/CCM.0000000000000852. PMID 25574794
- [Background] Jox RJ, Krebs M, Fegg M, Reiter-Theil S, Frey L, Eisenmenger W, Borasio GD. Limiting life-sustaining treatment in German intensive care units: a multiprofessional survey. J Crit Care. 2010 Sep;25(3):413-9. doi: 10.1016/j.jcrc.2009.06.012. Epub 2009 Aug 13. PMID 19682847
- [Background] Filip X, Filip C. Can the conformation of flexible hydroxyl groups be constrained by simple NMR crystallography approaches? The case of the quercetin solid forms. Solid State Nucl Magn Reson. 2015 Feb;65:21-8. doi: 10.1016/j.ssnmr.2014.10.006. Epub 2014 Nov 4. PMID 25465481
- [Background] Garcia AKA, Furuya RK, Conchon MF, Rossetto EG, Dantas RAS, Fonseca LF. Menthol chewing gum on preoperative thirst management: randomized clinical trial. Rev Lat Am Enfermagem. 2019 Oct 7;27:e3180. doi: 10.1590/1518-8345.3070.3180. eCollection 2019. PMID 31596415
- [Background] Woo K, Hill R, LeBlanc K, Percival SL, Schultz G, Weir D, Swanson T, Mayer DO. Effect of a surfactant-based gel on patient quality of life. J Wound Care. 2018 Oct 2;27(10):664-678. doi: 10.12968/jowc.2018.27.10.664. PMID 30332359
- [Background] Saha S, Bose R, Chakraborty S, Ain R. Tipping the balance toward stemness in trophoblast: Metabolic programming by Cox6B2. FASEB J. 2022 Nov;36(11):e22600. doi: 10.1096/fj.202200703RR. PMID 36250984
- [Background] Demerouti E, Bakker AB, Nachreiner F, Schaufeli WB. A model of burnout and life satisfaction amongst nurses. J Adv Nurs. 2000 Aug;32(2):454-64. doi: 10.1046/j.1365-2648.2000.01496.x. PMID 10964195
- [Background] Roe KL, Barbeau KA. Uptake mechanisms for inorganic iron and ferric citrate in Trichodesmium erythraeum IMS101. Metallomics. 2014 Nov;6(11):2042-51. doi: 10.1039/c4mt00026a. PMID 25222699
- [Background] Clark D, Baur N, Clelland D, Garralda E, Lopez-Fidalgo J, Connor S, Centeno C. Mapping Levels of Palliative Care Development in 198 Countries: The Situation in 2017. J Pain Symptom Manage. 2020 Apr;59(4):794-807.e4. doi: 10.1016/j.jpainsymman.2019.11.009. Epub 2019 Nov 22. PMID 31760142
- [Background] Epstein RL. Antitrust aspects of the future health planning. Issues Health Care. 1981;2(1):36-41. No abstract available. PMID 10253126
- [Background] Angus DC, Barnato AE, Linde-Zwirble WT, Weissfeld LA, Watson RS, Rickert T, Rubenfeld GD; Robert Wood Johnson Foundation ICU End-Of-Life Peer Group. Use of intensive care at the end of life in the United States: an epidemiologic study. Crit Care Med. 2004 Mar;32(3):638-43. doi: 10.1097/01.ccm.0000114816.62331.08. PMID 15090940
- [Background] Serafim Junior V, Fernandes GMM, Oliveira-Cucolo JG, Pavarino EC, Goloni-Bertollo EM. Role of Tropomyosin-related kinase B receptor and brain-derived neurotrophic factor in cancer. Cytokine. 2020 Dec;136:155270. doi: 10.1016/j.cyto.2020.155270. Epub 2020 Sep 7. PMID 32911446